CLINICAL TRIAL: NCT05488054
Title: Use of a Wearable Muscle Oxygen Saturation Sensor in the Rehabilitation of High-School and Collegiate Athletes Recovering From Arthroscopic Hip and Knee Surgery
Brief Title: Muscle O2 Saturation and Hemoglobin Levels During Rehabilitation From Arthroscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, James E Voos, MD, Chairman, Department of Orthopaedic Surgery, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191389
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: ACL Injury; Hip Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Hip Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Patients will be enrolled in one of two arms: surgical patients undergoing physical therapy or healthy volunteers. Data from patients including O2 and hemoglobin levels in injured tissue will be collected to determine safe return to sport.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Healthy Individuals (Experimental): Healthy control patients with no history of knee or hip surgery for comparison of baseline values
  Interventions: Procedure: Monitored Work-out; Device: Moxy Oxygen Sensor Device
- Surgical Patients (Experimental): Patients who have undergone arthroscopic ACL surgery or arthroscopic hip surgery and are undergoing physical therapy for return to sport
  Interventions: Procedure: Physical Therapy; Device: Moxy Oxygen Sensor Device

INTERVENTIONS:
Procedure: Physical Therapy — Patients will undergo physical therapy following surgical intervention
  Arms: Surgical Patients
Procedure: Monitored Work-out — Healthy volunteers will undergo a monitored workout for comparison of data
  Arms: Healthy Individuals
Device: Moxy Oxygen Sensor Device — Individuals will wear a Moxy sensor device during workouts to monitor oxygen and hemoglobin levels in their muscles

SUMMARY:
This study will utilize the Moxy wearable sensor to measure muscle oxygen saturation levels in athletes following lower extremity surgery (ACL or Hip arthroscopy) to evaluate their Return-to-Play. The acquired data will complement current protocols utilized by Dr. Voos and Dr. Salata in this regard and will add quantifiable evidence to enable a robust measurement of the surgical limb versus non-surgical limb.

DETAILED DESCRIPTION:
Patients with a diagnosis of ACL tear or hip pathology will undergo surgery. Following surgery, patients will report to clinic for scheduled physical therapy per their institution's injury-specific physical therapy protocol. At set time points (6-week, 12-week, 6 months, and 9 months) during their recovery, patients will be assessed for muscle oxygen saturation and hemoglobin levels with the Moxy sensor. This sensor is a non-invasive device placed over the rectus femoris to monitor oxygen and hemoglobin levels. The patient will then follow the therapy as instructed by the physical therapist and perform the protocol-specific exercises with the sensor in place. The measured parameters will be recorded and stored per patient.

The injured patients will be compared to healthy control patients undergoing a similar one-hour exercise session while wearing the Moxy sensor for comparison of results.

The goal of this study is to use the data obtained from the Moxy sensor device to further predict recovery of function in muscles supporting injured soft tissues to determine safe return to sport.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Patients age 14 to 30 years
* Patients with ACL injury requiring surgical correction
* Patients undergoing arthroscopic hip surgery
* Healthy individuals with no history of ACL, arthroscopic knee or arthroscopic hip surgery

Exclusion Criteria:

* Patients below 14 years or above 30 years
* Non-English-speaking subjects
* Pregnant individuals

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 226 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in O2 Saturation levels as measured by Moxy Sensor device | 6 months, 9 months, 12 months (once for healthy individuals)
Changes in hemoglobin levels as measured by Moxy Sensor device | 6 months, 9 months, 12 months (once for healthy individuals)

CONTACTS AND LOCATIONS:
Overall Officials: James Voos, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Sunita Mengers, MD, Study Director — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - University Hospitals Physical Therapy, Avon, Ohio
  - University Hospitals Cleveland Medial Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No